CLINICAL TRIAL: NCT01068652
Title: Effect of 50-week Treatment With Stepwise Insulin Intensification of Basal-bolus Insulin Analogues (Insulin Detemir and Aspart) or Biphasic Insulin Aspart 30 (NovoMix 30) All in Combination With Fixed Dose of Metformin on Glycaemic Control (Measured as HbA1c) in Subjects With Type 2 Diabetes. Open Labelled, Randomized, Two-arm, Parallel Group, Multi-centre, Multi-national Trial
Brief Title: Effect of Different Insulin Administrations, All in Combination With Metformin, on Glycaemic Control in Subjects With Type 2 Diabetes Inadequately Controlled by Oral Anti-diabetic Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INS-3782; U1111-1112-6407 (Other: WHO)
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart; insulin aspart, insulin aspart protamine drug combination 30:70; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Detemir + Met (Active Comparator): Individually adjusted insulin detemir (Detemir) was given subcutaneoulsy (s.c.) at bedtime in the thigh at an initial dose of 0.1 U/kg once daily for 50 weeks in combination with 1000-2000 mg/day metformin (Met). Pending evaluation of HbA1c every 3 months, individually adjusted insulin aspart was added to the insulin detemir treatment (up to three doses daily for maximum 36 weeks, injected s.c. [under the skin]) if treatment target of HbA1c below 7.0% was not reached.
  Interventions: Drug: insulin detemir; Drug: insulin aspart; Drug: metformin
- BIAsp 30 + Met (Active Comparator): Individually adjusted biphasic insulin aspart 30 (BIAsp 30) was given subcutaneously (s.c.) in the abdomen at dinner at an initial dose of 0.1 U/kg once daily for 50 weeks in combination with 1000-2000 mg/day metformin (Met). Pending evaluation of HbA1c every 3 months, the dose was intensified up to 3 doses daily, injected s.c. (under the skin) if treatment target of HbA1c below 7.0% was not reached.
  Interventions: Drug: biphasic insulin aspart 30; Drug: metformin

INTERVENTIONS:
Drug: insulin detemir — Initial dose of 0.1 U/kg once daily, injected s.c. (under the skin).
  Arms: Detemir + Met
Drug: insulin aspart — Pending evaluation of HbA1c every 3 months, insulin aspart was added to the insulin detemir treatment (up to three does daily, injected s.c. (under the skin)
  Arms: Detemir + Met
Drug: biphasic insulin aspart 30 — Initial dose of 0.1 U/kg once daily, injected s.c. (under the skin). Pending evaluation of HbA1c every 3 months, the dose will intensified up to 3 doses daily
  Arms: BIAsp 30 + Met
Drug: metformin — 1000-2000 mg/day in combination with insulin treatment

SUMMARY:
This trial is conducted in Africa. The aim of this clinical trial is to investigate the effect of 50 weeks of treatment with different intensified insulin administrations (all in combination with a fixed dose of metformin) on blood sugar control in subjects with type 2 diabetes inadequately controlled by oral anti-diabetic drugs (OADs).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject)
* Diagnosed type 2 diabetes (WHO 1999 criteria)
* Currently treated with suboptimal daily dose of OADs (mono or combination therapy) for at least 6 months
* Male or female age at least 18 years old
* HbA1c at least 7.0 % and maximum 11.0% for subjects treated with metformin mono-therapy, or maximum 10% for subjects treated with OAD combination therapy
* BMI maximum 40 kg/m^2
* Able and willing to perform self-monitoring of plasma glucose according to the protocol and to keep a diary
* Able and willing to be treated with up to 4 insulin injections per day

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Previous participation in this trial. Participation is defined as randomisation
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* Participated in another clinical trial and received an investigational drug within the last weeks prior to the present trial
* Impaired hepatic function defined as alanine aminotransferase (ALT) or alkaline phosphatase (ALP) at least 2.5 times upper referenced limit
* Impaired renal function defined as serum-creatinine at least 1.3 mg/dL (at least 115 mmol/L) for males and at least 1.2 mg/dL (at least 106 mmol/L) for females
* Subject has a clinically significant, active (or over the past 12 months) cardiovascular history (including a history of myocardial infarction (MI), arrhythmias or conduction delays on ECG, unstable angina, or decompensated heart failure (New York Heart Association class III and IV)
* Severe uncontrolled treated or untreated hypertension (sitting systolic blood pressure at least 180 mmHg or sitting diastolic blood pressure at least 100 mmHg)
* Proliferative retinopathy or macular oedema requiring acute treatment
* Metformin contraindications according to the package insert
* Current treatment with systemic corticosteroids
* Subject has a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering study drug to the subject
* Current addiction to alcohol or other addictive substances as determined by the Investigator
* Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation in the study or use of the glucose monitor
* History of hypoglycaemic unawareness and/or two or more severe hypoglycaemic episodes in the past year as judged by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2010-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (17):
- Algeria (6):
  - Novo Nordisk Investigational Site, Ain Témouchent
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Constantine
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sétif
  - Novo Nordisk Investigational Site, Sidi Bel Abbes
- Novo Nordisk Investigational Site, Alexandria, Egypt
- Novo Nordisk Investigational Site, Casablanca, Morocco
- South Africa (8):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Vaderbijlpark, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Kimberly, Northern Cape
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
  - Novo Nordisk Investigational Site, Sandton
- Novo Nordisk Investigational Site, Tunisia, Tunisia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 23 sites in 4 countries: Egypt (1), Algeria (9), Tunisia (4) and South Africa (9). The trial consisted of two weeks of screening, three weeks of run-in, and 50 weeks of treatment.
Period: Overall Study
Arm/Group | Detemir + Met | BIAsp 30 + Met
Started | 200 | 203
Completed | 182 | 188
Not Completed | 18 | 15
Not completed — Adverse Event | 4 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Protocol Violation | 3 | 6
Not completed — Withdrawal criteria | 1 | 2
Not completed — Patient was not eligible | 1 | 0
Not completed — Unclassified | 7 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Detemir + Met | BIAsp 30 + Met | Total
Number analyzed (Participants) | 200 | 203 | 403
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (9.0) | 52.6 (10.1) | 52.8 (9.6)
Gender [Count of Participants; unit: Participants]
  Female | 113 | 128 | 241
  Male | 87 | 75 | 162
Race/Ethnicity, Customized [Number; unit: participants]
  White | 54 | 58 | 112
  Black or African American | 18 | 11 | 29
  Asian | 16 | 21 | 37
  Other | 112 | 113 | 225
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.6 (1.1) | 8.7 (1.1) | 8.7 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin (HbA1c)
Description: Estimated mean difference in HbA1c after 50 weeks of treatment
Time Frame: Week 50
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF). For 20 subjects, HbA1c values were missing.
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 191 | 192
percentage of glycosylated haemoglobin | 7.34 (0.13) | 7.23 (0.12)
Statistical Analysis 1: Comparison: Detemir + Met vs BIAsp 30 + Met; To investigate the effect of different treatments, an analysis of covariance (ANCOVA) model was used to analyse HbA1c at week 50 with treatment group (2 categories: insulin detemir and aspart; BIAsp 30), country and pre-trial OAD(s) treatment (one OAD vs. more OADs) as factors and HbA1c at baseline (week 0) as a covariate. The treatment difference was estimated and a 95% confidence interval (CI) for the difference was calculated; Test type: Non-Inferiority or Equivalence — The treatment comparison was based on a non-inferiority criterion and the following hypotheses were tested: H0: μDetemir - μBIAsp 30 ≥0.4% against the alternative hypothesis (Detemir non-inferior to BIAsp 30) HA: μDetemir - μBIAsp 30 <0.4% where μBIAsp 30 and μDetemir are the mean HbA1c after 50 weeks of treatment with the two treatment regimens; p = 0.3406, ANCOVA; Mean Difference (Final Values) = 0.11, 95% CI [-0.12 to 0.34]

2. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) After 14 Weeks of Treatment
Description: Observed mean change from baseline in HbA1c at Week 14 (visit 11)
Time Frame: Week 0, Week 14
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF). For 20 subjects, values for change in HbA1c were missing.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 191 | 192
percentage of glycosylated haemoglobin | -0.18 (1.16) | -0.64 (1.12)

3. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) After 26 Weeks of Treatment
Description: Observed mean change in from baseline in HbA1c at Week 26 (visit 18)
Time Frame: Week 0, Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 191 | 192
percentage of glycosylated haemoglobin | -1.05 (1.05) | -1.30 (1.28)

4. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) After 38 Weeks of Treatment
Description: Observed mean change from baseline in HbA1c at Week 38 (visit 25)
Time Frame: Week 0, Week 38
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 191 | 192
percentage of glycosylated haemoglobin | -1.35 (1.16) | -1.56 (1.39)

5. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c) at Week 50
Description: Observed mean change from baseline in HbA1c at Week 50 (visit 32)
Time Frame: Week 0, Week 50
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 191 | 192
percentage of glycosylated haemoglobin | -1.16 (1.33) | -1.34 (1.40)

6. Secondary Outcome: Number of Subjects Achieving Glycosylated Haemoglobin (HbA1c) Below 7.0% After 14 Weeks of Treatment
Description: Number of subjects achieving HbA1c below 7.0% after 14 weeks of treatment (visit 11)
Time Frame: Week 14
Population: Full Analysis Set (FAS) includes all randomised subjects. For 20 subjects, values were missing.
Measure: Number; unit: Subjects
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 191 | 192
Subjects | 15 | 26

7. Secondary Outcome: Number of Subjects Achieving Glycosylated Haemoglobin (HbA1c) Below 7.0% After 26 Weeks of Treatment
Description: Number of subjects achieving HbA1c below 7.0% after 26 weeks of treatment (visit 18)
Time Frame: Week 26
Population: Full Analysis Set (FAS) includes all randomised subjects. For 29 subjects, values were missing.
Measure: Number; unit: Subjects
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 185 | 189
Subjects | 67 | 77

8. Secondary Outcome: Number of Subjects Achieving Glycosylated Haemoglobin (HbA1c) Below 7.0% After 38 Weeks of Treatment
Description: Number of subjects achieving HbA1c below 7.0% after 38 weeks of treatment (visit 25)
Time Frame: Week 38
Population: Full Analysis Set (FAS) includes all randomised subjects. For 31 subjects, values were missing.
Measure: Number; unit: Subjects
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 184 | 188
Subjects | 84 | 103

9. Secondary Outcome: Number of Subjects Achieving Glycosylated Haemoglobin (HbA1c) Below 7.0% After 50 Weeks of Treatment
Description: Number of subjects achieving HbA1c below 7.0% after 50 weeks of treatment (visit 32)
Time Frame: Week 50
Population: Full Analysis Set (FAS) includes all randomised subjects. For 35 subjects, values were missing.
Measure: Number; unit: Subjects
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 181 | 187
Subjects | 73 | 84

10. Secondary Outcome: Mean of Prandial Plasma Glucose (PG) Increment After 14 Weeks of Treatment
Description: Observed overall mean of PG increment after 14 weeks of treatment (Visit 11). Mean PG Increment was calculated using the average of difference between the Post Prandial and Pre Prandial Glucose values {ie .average of (Post Breakfast - Pre Breakfast), (Post Lunch - Pre Lunch) and (Post Dinner - Pre Dinner)}
Time Frame: Week 14
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF). For 28 subjects, PG (mg/dL) increment values were missing at all evaluations.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 188 | 187
mg/dL | 43.19 (33.64) | 32.61 (31.99)

11. Secondary Outcome: Mean of Prandial Plasma Glucose (PG) Increment After 26 Weeks of Treatment
Description: Observed overall mean of PG increment after 26 weeks of treatment (visit 18). Mean PG Increment was calculated using the average of difference between the Post Prandial and Pre Prandial Glucose values {ie .average of (Post Breakfast - Pre Breakfast), (Post Lunch - Pre Lunch) and (Post Dinner - Pre Dinner)}
Time Frame: Week 26
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF). For 19 subjects, PG (mg/dL) increment values were missing at all evaluations.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 192 | 192
mg/dL | 32.95 (30.25) | 31.71 (27.86)

12. Secondary Outcome: Mean of Prandial Plasma Glucose (PG) Increment After 38 Weeks of Treatment
Description: Observed overall mean of PG increment after 38 weeks of treatment (visit 25). Mean PG Increment was calculated using the average of difference between the Post Prandial and Pre Prandial Glucose values {ie .average of (Post Breakfast - Pre Breakfast), (Post Lunch - Pre Lunch) and (Post Dinner - Pre Dinner)}.
Time Frame: Week 38
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 192 | 192
mg/dL | 25.44 (27.95) | 28.32 (30.69)

13. Secondary Outcome: Mean of Prandial Plasma Glucose (PG) Increment After 50 Weeks of Treatment
Description: Observed overall mean of PG increment after 50 weeks of treatment (visit 32). Mean PG Increment was calculated using the average of difference between the Post Prandial and Pre Prandial Glucose values {ie .average of (Post Breakfast - Pre Breakfast), (Post Lunch - Pre Lunch) and (Post Dinner - Pre Dinner)}.
Time Frame: Week 50
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 192 | 192
mg/dL | 22.45 (25.50) | 23.66 (28.91)

14. Secondary Outcome: Mean of 8-point Plasma Glucose (PG) Profile After 14 Weeks of Treatment
Description: Observed overall mean of 8-point PG profile after 14 weeks of treatment (visit 11)
Time Frame: Week 14
Population: Full analysis set (FAS) includes all randomised subjects and missing data is imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 200 | 203
mg/dL
  Before Breakfast (n=193, 194) | 136.44 (42.86) | 128.31 (33.58)
  120 min After Breakfast (n=187, 184) | 181.89 (54.42) | 176.31 (44.50)
  Before Lunch (n=192, 193) | 157.61 (53.43) | 156.12 (51.57)
  120 min After Lunch (n=186, 185) | 199.40 (64.38) | 199.75 (59.04)
  Before Dinner (n=191, 192) | 169.69 (54.91) | 168.09 (59.58)
  120 min After Dinner (n=183, 185) | 212.23 (61.45) | 173.95 (54.86)
  Bedtime (n=187, 192) | 200.15 (60.83) | 156.65 (50.65)
  At 2 AM - 3 AM (n=172, 177) | 158.69 (50.06) | 139.93 (43.39)

15. Secondary Outcome: Mean of 8-point Plasma Glucose (PG) Profile After 26 Weeks of Treatment
Description: Observed overall mean of 8-point PG profile after 26 weeks of treatment (visit 18)
Time Frame: Week 26
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 200 | 203
mg/dL
  Before Breakfast (n=193, 194) | 116.57 (34.40) | 115.79 (27.23)
  120 min After Breakfast (n=191, 191) | 163.52 (50.02) | 153.85 (42.68)
  Before Lunch (n=193, 194) | 140.97 (49.96) | 131.27 (42.85)
  120 min After Lunch (n=191, 191) | 166.00 (57.15) | 178.92 (51.14)
  Before Dinner (n=192, 194) | 147.58 (48.90) | 143.29 (45.50)
  120 min After Dinner (n=188, 191) | 172.21 (57.34) | 152.44 (45.53)
  Bedtime (n=190, 194) | 164.70 (63.68) | 140.39 (42.71)
  At 2 AM - 3 AM (n=181, 187) | 133.59 (47.54) | 123.29 (35.16)

16. Secondary Outcome: Mean of 8-point Plasma Glucose (PG) Profile After 38 Weeks of Treatment
Description: Observed overall mean of 8-point PG profile after 38 weeks of treatment (visit 25)
Time Frame: Week 38
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 200 | 203
mg/dL
  Before Breakfast (n=193, 194) | 110.14 (30.64) | 110.86 (27.11)
  120 min After Breakfast (n=191, 192) | 146.70 (44.11) | 139.38 (42.74)
  Before Lunch (n=193, 194) | 130.63 (42.17) | 118.30 (40.28)
  120 min After Lunch (n=191, 192) | 145.91 (51.38) | 158.45 (47.70)
  Before Dinner (n=193, 194) | 132.26 (41.90) | 129.10 (43.84)
  120 min After Dinner (n=192,192) | 155.47 (49.09) | 142.82 (50.47)
  Bedtime (n=193, 194) | 146.37 (51.58) | 132.45 (43.54)
  At 2 AM - 3 AM (n=187, 190) | 124.57 (42.11) | 117.42 (35.60)

17. Secondary Outcome: Mean of 8-point Plasma Glucose (PG) Profile After 50 Weeks of Treatment
Description: Observed overall mean of 8-point PG profile after 50 weeks of treatment (visit 32)
Time Frame: Week 50
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Detemir + Met | BIAsp 30 + Met
Number analyzed (Participants) | 200 | 203
mg/dL
  Before Breakfast (n=193, 194) | 108.78 (31.10) | 110.76 (22.08)
  120 min After Breakfast (n=191, 192) | 140.05 (40.98) | 132.45 (35.55)
  Before Lunch (n=193, 194) | 120.43 (37.62) | 115.02 (36.20)
  120 min After Lunch (n=191, 192) | 139.48 (49.03) | 149.90 (44.32)
  Before Dinner (n=193, 194) | 128.28 (40.63) | 126.76 (40.16)
  120 min After Dinner (n=192, 192) | 144.19 (49.24) | 138.08 (42.11)
  Bedtime (n=193, 194) | 137.13 (51.18) | 130.10 (43.08)
  At 2 AM - 3 AM (n=187, 190) | 118.60 (40.65) | 113.14 (35.21)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 0-50 weeks + 2 weeks follow-up
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator
Arm/Group | Detemir + Met | BIAsp 30 + Met
Serious Adverse Events (participants affected / at risk) | 13/200 | 7/203
Other Adverse Events (participants affected / at risk) | 75/200 | 78/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Detemir + Met (N=200) | BIAsp 30 + Met (N=203)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ECG signs of myocardial ischaemia (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Detemir + Met (N=200) | BIAsp 30 + Met (N=203)
Abdominal pain upper (Gastrointestinal disorders) | 16 (17) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 13 (15) | 15 (20)
Influenza (Infections and infestations) | 15 (20) | 17 (20)
Urinary tract infection (Infections and infestations) | 10 (11) | 11 (13)
Headache (Nervous system disorders) | 13 (18) | 12 (12)
Hypertension (Vascular disorders) | 8 (8) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.